CLINICAL TRIAL: NCT04877990
Title: An Open-label, Multi-center Extension Study to Evaluate the Long-term Safety and Efficacy of Deucravacitinib in Participants With Moderate to Severe Crohn's Disease or Moderate to Severe Ulcerative Colitis
Brief Title: A Study to Evaluate the Long-term Safety and Efficacy of Deucravacitinib in Participants With Crohn's Disease or Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM011-077; 2020-004461-40 (EudraCT Number); U1111-1258-3838 (Registry Identifier: WHO)
Record Dates: First submitted 2021-05-04; First posted 2021-05-07 (Actual); Results first posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-08

CONDITIONS: Crohn Disease; Ulcerative Colitis
Keywords: BMS-986165; Crohn Colitis; Crohn Disease; Crohn Iliocolitis; Inflammatory Bowel Disease; Ulcerative Colitis; Deucravacitinib
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — deucravacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Long-Term Extension Rollover Study: Deucravacitinib (Experimental)
  Interventions: Drug: Deucravacitinib

INTERVENTIONS:
Drug: Deucravacitinib — Specified dose on specified days

SUMMARY:
The purpose of this study is to evaluate the long-term safety and efficacy of Deucravacitinib in participants who have previously been enrolled in a Deucravacitinib Phase 2 study for moderate to severe Crohn's disease or moderate to severe Ulcerative Colitis.

ELIGIBILITY:
Inclusion Criteria:

• Previously completed open-label extension treatment in one of the parent Crohn's disease or ulcerative colitis studies

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Current colonic adenomas or dysplasia diagnosed at the endoscopy performed at the end of treatment visit of the parent study or past confirmed colonic dysplasia in the parent study that has not been eradicated

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (43):
- United States (10):
  - Local Institution - 0036, Shreveport, Louisiana
  - Local Institution - 0002, Wyoming, Michigan
  - Local Institution - 0037, Jackson, Mississippi
  - Local Institution - 0041, Cleveland, Ohio
  - Local Institution - 0038, Pittsburgh, Pennsylvania
  - Local Institution - 0066, Charleston, South Carolina
  - Local Institution - 0053, Garland, Texas
  - Local Institution - 0056, San Antonio, Texas
  - Local Institution - 0049, Tyler, Texas
  - Local Institution - 0055, Richmond, Virginia
- Local Institution - 0013, Ballarat, Victoria, Australia
- Local Institution - 0050, Vaughan, Ontario, Canada
- China (2):
  - Local Institution - 0030, Guangzhou, Guangdong
  - Local Institution - 0029, Guangzhou, Guangdong
- Local Institution - 0012, Kiel, Germany
- Hungary (2):
  - Local Institution - 0062, Budapest
  - Local Institution - 0023, Budapest
- Italy (2):
  - Humanitas, Rozzano, Lombardy
  - Fondazione Irccs - Policlinico San Matteo, Pavia
- Japan (5):
  - Local Institution - 0063, Hirosaki, Aomori
  - Local Institution - 0047, Sagamihara, Kanagawa
  - Local Institution - 0027, Saga, Saga-ken
  - Local Institution - 0026, Bunkyo-ku, Tokyo
  - Local Institution - 0044, Minato-ku, Tokyo
- Local Institution - 0060, Amsterdam, North Holland, Netherlands
- Poland (11):
  - Local Institution - 0046, Nowy Targ, Lesser Poland Voivodeship
  - Local Institution - 0061, Tychy, Silesian Voivodeship
  - Local Institution - 0022, Bydgoszcz
  - Local Institution - 0003, Bydgoszcz
  - Local Institution - 0001, Krakow
  - Local Institution - 0028, Sopot
  - Local Institution - 0025, Szczecin
  - Local Institution - 0035, Warsaw
  - Local Institution - 0048, Warsaw
  - Local Institution - 0004, Warsaw
  - Local Institution - 0018, Wroclaw
- Local Institution - 0054, Santa Maria da Feira, Portugal
- Local Institution, Bucharest, Romania
- Russia (2):
  - Local Institution, Irkutsk
  - Local Institution, Saint Petersburg
- Local Institution - 0045, Fuenlabrada, Madrid, Spain
- Local Institution - 0064, Taipei, Taiwan
- Local Institution - 0034, Morriston, United Kingdom

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Crohn's Disease; Ulcerative Colitis: Deucravacitinib (BMS-986165) 6 mg twice daily (BID)
Period: Pre-treatment
Arm/Group | Crohn's Disease | Ulcerative Colitis
Started (Started=Randomized) | 26 | 41
Completed (Completed=Treated) | 24 | 41
Not Completed | 2 | 0
Period: Treatment
Arm/Group | Crohn's Disease | Ulcerative Colitis
Started | 24 | 41
Completed | 0 | 0
Not Completed | 24 | 41
Not completed — Other reasons | 3 | 1
Not completed — Administrative reasons by sponsor | 17 | 33
Not completed — Withdrawal by Subject | 2 | 6
Not completed — Adverse Event | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Crohn's Disease | Ulcerative Colitis | Total
Number analyzed (Participants) | 26 | 41 | 67
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.7 (14.08) | 44.3 (15.70) | 42.2 (15.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 19 | 29
  Male | 16 | 22 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 21 | 35 | 56
  Unknown or Not Reported | 5 | 5 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 21 | 38 | 59
  Black or African American | 1 | 0 | 1
  Asian | 2 | 0 | 2
  American Indian or Alaska Native | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Other | 0 | 0 | 0
  Asian Indian | 0 | 0 | 0
  Chinese | 2 | 0 | 2
  Japanese | 0 | 3 | 3
  Asian Other | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: Number of participants experiencing AEs, SAEs, AEs leading to study discontinuation, and AEs of interest (AEIs). An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment. SAEs is any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires inpatient hospitalization; results significant disability; or is a congenital anomaly/birth defect. TEAEs are defined as AEs with an onset date on or after the first dose of study treatment up to 30 days after the last dose of study treatment in the study, or if a pre-existing condition worsens in severity or becomes serious after receiving the first dose of study treatment
Time Frame: From first dose to 30 days post last dose (Up to 110 weeks)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Crohn's Disease | Ulcerative Colitis
Number analyzed (Participants) | 24 | 41
Participants
  TEAEs | 18 | 19
  TESAEs | 2 | 2
  TEAEs leading to study discontinuation | 1 | 1
  AEs of Interest - Skin-related events | 0 | 2
  AEs of Interest - Creatine Kinase events | 2 | 3

2. Primary Outcome: Number of Participants With Laboratory Abnormalities
Description: Number of participants experiencing abnormalities in laboratory testing including chemistry, hematology, and renal.
Time Frame: From first dose to 30 days post last dose (Up to 110 weeks)
Population: All treated participants with laboratory measurements
Measure: Count of Participants; unit: Participants
Arm/Group | Crohn's Disease | Ulcerative Colitis
Number analyzed (Participants) | 23 | 41
Participants
  Sodium < 130 or > 150 MEQ/L (MMOL/L) | 0 | 0
  Potassium < 3 or > 5.5 MEQ/L (MMOL/L) | 0 | 1
  Calcium > 12.5 MG/DL | 0 | 0
  Fasting Serum Glucose < 50 MG/DL or > 250 MG/DL: number analyzed (Participants) | 16 | 28
  Fasting Serum Glucose < 50 MG/DL or > 250 MG/DL | 0 | 0
  Albumin < 2.0 G/DL | 0 | 0
  Creatine Kinase > 10xupper limit of normal | 0 | 0
  Hemoglobin < 7.0 G/DL or > 30% reduction from baseline: number analyzed (Participants) | 23 | 40
  Hemoglobin < 7.0 G/DL or > 30% reduction from baseline | 0 | 0
  Hematocrit < 20% or 30% reduction from baseline: number analyzed (Participants) | 23 | 40
  Hematocrit < 20% or 30% reduction from baseline | 0 | 0
  White Blood Cell Count < 1.5 x 10^9/L or > 35 x 10^9/L: number analyzed (Participants) | 23 | 40
  White Blood Cell Count < 1.5 x 10^9/L or > 35 x 10^9/L | 0 | 0
  Lymphocyte Count < 0.5 x 10^9/L: number analyzed (Participants) | 23 | 40
  Lymphocyte Count < 0.5 x 10^9/L | 0 | 0
  Neutrophil Count < 0.75 x 10^9/L: number analyzed (Participants) | 23 | 40
  Neutrophil Count < 0.75 x 10^9/L | 0 | 0
  Platelet Count < 75 x 10^9/L or > 999 x 10^9/L: number analyzed (Participants) | 23 | 40
  Platelet Count < 75 x 10^9/L or > 999 x 10^9/L | 0 | 0
  Serum Creatinine Increase > 50% and > 44.2 UMOL/L | 0 | 0

3. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities
Time Frame: From first dose to 30 days post last dose (Up to 110 weeks)
Population: All treated participants with ECG measurements
Measure: Count of Participants; unit: Participants
Arm/Group | Crohn's Disease | Ulcerative Colitis
Number analyzed (Participants) | 24 | 41
Participants
  QTCF (MSEC) 450 - < 480 | 1 | 0
  QTCF (MSEC) 480 - < 500 | 0 | 1
  QTCF (MSEC) >= 500 | 0 | 0
  30 < CHANGE FROM IM011077 STUDY BASELINE <= 60 MSEC | 3 | 0
  CHANGE FROM IM011077 STUDY BASELINE > 60 MSEC | 3 | 5
  PRAG (MSEC) P WAVE AND R WAVE (PR) INTERVAL >= 240 MSEC | 0 | 0
  QRSAG(MSEC) QRS INTERVAL >= 200 MSEC | 0 | 0

4. Primary Outcome: Number of Participants With Vital Signs Abnormalities
Time Frame: From first dose to 30 days post last dose (Up to 110 weeks)
Population: All treated participants with vital signs measurements
Measure: Count of Participants; unit: Participants
Arm/Group | Crohn's Disease | Ulcerative Colitis
Number analyzed (Participants) | 24 | 41
Participants
  HEART RATE (BEATS/MIN): VALUE > 100 AND CHANGE FROM IM011077 STUDY BASELINE > 30 | 1 | 1
  HEART RATE (BEATS/MIN): VALUE < 55 AND CHANGE FROM IM011077 STUDY BASELINE < -15 | 1 | 0
  SYSTOLIC BLOOD PRESSURE (MMHG): VALUE > 140 AND CHANGE FROM IM011077 STUDY BASELINE > 20 | 3 | 5
  SYSTOLIC BLOOD PRESSURE (MMHG): VALUE < 90 AND CHANGE FROM IM011077 STUDY BASELINE < -20 | 0 | 0
  DIASTOLIC BLOOD PRESSURE (MMHG): VALUE > 90 AND CHANGE FROM IM011077 STUDY BASELINE > 10 | 3 | 5
  DIASTOLIC BLOOD PRESSURE (MMHG): VALUE < 55 AND CHANGE FROM IM011077 STUDY BASELINE < -10 | 0 | 0

5. Primary Outcome: Change From Baseline in Laboratory Parameters
Description: Change from baseline in laboratory parameters including lipid profile, chemistry liver function, chemistry (other), and chemistry renal function
Time Frame: Baseline, Week 12, Week 108
Population: All treated participants with baseline and post baseline measurements at pre-specified time points
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Crohn's Disease | Ulcerative Colitis
Number analyzed (Participants) | 23 | 38
mg/dL
  Cholesterol, Fasting Week 12: number analyzed (Participants) | 5 | 6
  Cholesterol, Fasting Week 12 | 10.20 (7.207) | -9.17 (4.629)
  Cholesterol, Fasting Week 108: number analyzed (Participants) | 1 | 0
  Cholesterol, Fasting Week 108 | -12.00 (NA) — insufficient number of participants with events |
  HDL Cholesterol, Fasting Week 12: number analyzed (Participants) | 4 | 6
  HDL Cholesterol, Fasting Week 12 | -0.75 (3.400) | -0.83 (2.626)
  HDL Cholesterol, Fasting Week 108: number analyzed (Participants) | 1 | 0
  HDL Cholesterol, Fasting Week 108 | 0.00 (NA) — insufficient number of participants with events |
  LDL Cholesterol, Fasting Week 12: number analyzed (Participants) | 4 | 6
  LDL Cholesterol, Fasting Week 12 | 4.75 (4.270) | -6.50 (4.689)
  LDL Cholesterol, Fasting Week 108: number analyzed (Participants) | 1 | 0
  LDL Cholesterol, Fasting Week 108 | 1.00 (NA) — insufficient number of participants with events |
  Triglycerides, Fasting Week 12: number analyzed (Participants) | 4 | 6
  Triglycerides, Fasting Week 12 | 2.3 (11.31) | 3.2 (4.78)
  Triglycerides, Fasting Week 108: number analyzed (Participants) | 1 | 0
  Triglycerides, Fasting Week 108 | -62.0 (NA) — insufficient number of participants with events |
  Bilirubin, Week 12: number analyzed (Participants) | 22 | 36
  Bilirubin, Week 12 | 0.0650 (0.05028) | 0.0043 (0.03566)
  Bilirubin, Week 108: number analyzed (Participants) | 2 | 0
  Bilirubin, Week 108 | -0.1000 (0.00000) |
  Glucose, Fasting Serum Week 12: number analyzed (Participants) | 4 | 5
  Glucose, Fasting Serum Week 12 | 1.75 (0.946) | 0.80 (1.114)
  Glucose, Fasting Serum Week 108: number analyzed (Participants) | 1 | 0
  Glucose, Fasting Serum Week 108 | 29.00 (NA) — insufficient number of participants with events |
  Calcium, Week 12 | 0.152 (0.0915) | 0.041 (0.0612)
  Calcium, Week 108: number analyzed (Participants) | 2 | 0
  Calcium, Week 108 | 0.350 (0.1500) |
  Creatinine, Week 12: number analyzed (Participants) | 23 | 37
  Creatinine, Week 12 | -0.008 (0.0182) | 0.004 (0.0153)
  Creatinine, Week 108: number analyzed (Participants) | 2 | 0
  Creatinine, Week 108 | 0.080 (0.0100) |
  Phosphate, Week 12: number analyzed (Participants) | 19 | 37
  Phosphate, Week 12 | 0.153 (0.0893) | 0.019 (0.1198)
  Phosphate, Week 108: number analyzed (Participants) | 2 | 0
  Phosphate, Week 108 | -0.150 (0.1500) |
  Urea Nitrogen, Week 12: number analyzed (Participants) | 13 | 28
  Urea Nitrogen, Week 12 | -0.269 (1.0631) | 0.511 (0.5902)
  Urea Nitrogen, Week 108: number analyzed (Participants) | 2 | 0
  Urea Nitrogen, Week 108 | 5.500 (0.5000) |

6. Primary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameters - ECG Mean Heart Rate
Description: Changes from IM011077 study baseline in electrocardiogram (ECG) parameters - ECG mean heart rate
Time Frame: Baseline, Week 48, Week 96
Population: All treated participants with baseline and post baseline measurements at pre-specified time points
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Crohn's Disease | Ulcerative Colitis
Number analyzed (Participants) | 9 | 17
beats/min
  ECG Mean Heart Rate, Week 48 | -1.4 (9.21) | 2.6 (12.76)
  ECG Mean Heart Rate, Week 96: number analyzed (Participants) | 3 | 1
  ECG Mean Heart Rate, Week 96 | -1.0 (11.27) | -1.0 (NA) — insufficient number of participants with events

7. Primary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameters
Description: Changes from IM011077 study baseline in electrocardiogram (ECG) parameters
Time Frame: Baseline, Week 48, Week 96
Population: All treated participants with baseline and post baseline measurements at pre-specified time points
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Crohn's Disease | Ulcerative Colitis
Number analyzed (Participants) | 9 | 16
msec
  PR Interval, Aggregate, Week 48: number analyzed (Participants) | 9 | 15
  PR Interval, Aggregate, Week 48 | 9.1 (20.62) | -2.4 (22.65)
  PR Interval, Aggregate, Week 96: number analyzed (Participants) | 3 | 1
  PR Interval, Aggregate, Week 96 | 14.7 (16.56) | -22.0 (NA) — insufficient number of participants with events
  QRS Duration, Aggregate, Week 48: number analyzed (Participants) | 9 | 15
  QRS Duration, Aggregate, Week 48 | -1.2 (8.47) | -0.9 (8.53)
  QRS Duration, Aggregate, Week 96: number analyzed (Participants) | 3 | 1
  QRS Duration, Aggregate, Week 96 | -9.3 (2.89) | 0.0 (NA) — insufficient number of participants with events
  QT Interval, Aggregate, Week 48 | 18.6 (30.33) | 7.6 (40.35)
  QT Interval, Aggregate, Week 96: number analyzed (Participants) | 3 | 1
  QT Interval, Aggregate, Week 96 | 27.0 (62.55) | 96.0 (NA) — insufficient number of participants with events
  QTcB Interval, Aggregate, Week 48: number analyzed (Participants) | 3 | 9
  QTcB Interval, Aggregate, Week 48 | -2.3 (21.78) | 7.7 (19.41)
  QTcB Interval, Aggregate, Week 96: number analyzed (Participants) | 0 | 0
  QTcF Interval, Aggregate, Week 48 | -20.6388 (197.49472) | 31.1621 (141.14597)
  QTcF Interval, Aggregate, Week 96: number analyzed (Participants) | 3 | 1
  QTcF Interval, Aggregate, Week 96 | -86.9797 (198.61888) | 101.0000 (NA) — insufficient number of participants with events

8. Primary Outcome: Change From Baseline in Vital Signs Parameters - Heart Rate
Description: Changes from IM011077 study baseline in vital signs parameters - heart rate
Time Frame: Baseline, Week 12, Week 108
Population: All treated participants with baseline and post baseline measurements at pre-specified time points
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Crohn's Disease | Ulcerative Colitis
Number analyzed (Participants) | 24 | 41
beats/min
  Heart Rate Week 12 | 3.6 (11.89) | 0.9 (10.71)
  Heart Rate Week 108: number analyzed (Participants) | 1 | 0
  Heart Rate Week 108 | 1.0 (NA) — insufficient number of participants with events |

9. Primary Outcome: Change From Baseline in Vital Signs Parameters
Description: Changes from IM011077 study baseline in vital signs parameters
Time Frame: Baseline, Week 12, Week 108
Population: All treated participants with baseline and post baseline measurements at pre-specified time points
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Crohn's Disease | Ulcerative Colitis
Number analyzed (Participants) | 24 | 41
mmHg
  Systolic Blood Pressure Week 12 | 3.8 (11.56) | 3.8 (13.62)
  Systolic Blood Pressure Week 108: number analyzed (Participants) | 1 | 0
  Systolic Blood Pressure Week 108 | 4.0 (NA) — insufficient number of participants with events |
  Diastolic Blood Pressure Week 12 | 0.3 (7.82) | -1.3 (7.38)
  Diastolic Blood Pressure Week 108: number analyzed (Participants) | 1 | 0
  Diastolic Blood Pressure Week 108 | 9.0 (NA) — insufficient number of participants with events |

ADVERSE EVENTS:
Time Frame: SAEs and AEs are assessed from first dose to 30 days post last dose (Up to 110 weeks). Participants were assessed for all-cause mortality from their first dose to study completion (Up to 120 weeks).
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication.
Arm/Group | CROHN'S DISEASE | ULCERATIVE COLITIS
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/41
Serious Adverse Events (participants affected / at risk) | 2/24 | 2/41
Other Adverse Events (participants affected / at risk) | 12/24 | 13/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CROHN'S DISEASE (N=24) | ULCERATIVE COLITIS (N=41)
Cardiac failure chronic (Cardiac disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
General physical health deterioration (General disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CROHN'S DISEASE (N=24) | ULCERATIVE COLITIS (N=41)
Colitis ulcerative (Gastrointestinal disorders) | 0 | 3
Mouth ulceration (Gastrointestinal disorders) | 2 | 1
Pyrexia (General disorders) | 2 | 1
COVID-19 (Infections and infestations) | 6 | 3
Nasopharyngitis (Infections and infestations) | 3 | 0
Pneumonia (Infections and infestations) | 3 | 0
Tonsillitis (Infections and infestations) | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 2 | 5
Depression (Psychiatric disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-04): https://cdn.clinicaltrials.gov/large-docs/90/NCT04877990/Prot_SAP_000.pdf